CLINICAL TRIAL: NCT02868528
Title: A Prospective Randomized Controlled Study of Preimplantation Genetic Screening With Next Generation Sequencing Technology on Advanced Age Women
Brief Title: A Study of Preimplantation Genetic Screening With Next Generation Sequencing Technology on Advanced Age Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KYXM-201603
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2020-03

CONDITIONS: Infertility
Keywords: advanced age women; blastocyst culture; PGS; live birth rate
MeSH Terms: conditions — Infertility

ARMS (2):
- PGS group (Experimental): After blastocyst culture, blastocyst embryo trophoblast biopsy will be performed and chromosome screening with NGS technology, at the same time, the blastocysts will be frozen, then the blastocysts with normal chromosome will be thawed and transferred.
  Interventions: Genetic: chromosome screening with NGS technology
- control group (No Intervention): After blastocyst culture, blastocysts will be transferred

INTERVENTIONS:
Genetic: chromosome screening with NGS technology
  Arms: PGS group

SUMMARY:
With the development of society, more and more aged pregnant women because of various reasons, their abnormality rate of egg chromosome was higher than that of young women, then the abnormality rate of embryo chromosome is higher too, so the pregnancy rate in aged women is lower, abortion rate is higher. In order to improve the pregnancy rate in aged women, cut down their abortion rate 、fetal birth with abnormal chromosome, and the risk of pregnancy termination after the prenatal diagnosis, reduce their pain of body and mind, the investigators will carry out this study. This is a prospective randomized controlled study of preimplantation genetic screening with Next generation sequencing technology. The embryos with more developmental potential and normal chromosomes should be selected. There is no related studies in Chinese. Most international research are limited to fluorescence in situ hybridization (FISH) technique, not on the embryo chromosome comprehensive screening. So there is no evidence of the effects of PGS on advanced age women.

This study is to compare the outcomes between the advanced age women with two methods respectively. After blastocyst culture, blastocysts will be transferred in the control group. In the Preimplantation Genetic Screening (PGS) group, blastocyst embryo trophoblast biopsy will be performed and chromosome screening with Next generation sequencing（NGS） technology, at the same time, the blastocysts will be frozen, then the blastocysts with normal chromosome will be thawed and transferred. The investigators expect that, in PGS group live birth rate 、cancellation rate and pregnancy rate are higher than in control group; abortion rate is lower than that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females, age ≥37 years ≤44 years
* Have given birth to a healthy baby
* Bilateral ovaries
* Antral follicle count(AFC)≥10,and Anti Mullerian Hormone (AMH)≥2.0 ng/ml

Exclusion Criteria:

* Endometriosis disease
* Intrauterine adhesions history; intrauterine membrane polyp, tuberculosis and inflammation,
* Uterine malformation, multiple uterine myoma, uterine intramural myoma >3cm, submucous myoma;
* Unprocessed hydrosalpinx
* Adverse reproductive history; greater than or equal to 2 times history of unexplained abortion
* Chromosomal abnormalities or other genetic disease
* Infertility caused by male factors, such as puncture testicular, SRT did not see the class A and class B sperm
* Without high quality embryos in past controlled ovarian hyperstimulation (COH)cycles.
* Patients with poor ovarian response, the standard of poor ovarian response accords with Bolognacriteria standard, that is at least meet 2 among the following 3:

  1. . Elder years (≥40 years) or have other known inherited or acquired risk factors that may reduce follicle.
  2. .History of cancellation of the cycles because of less than 3 follicular development, or history of egg number less than 4 after at least using Follicle-Stimulating Hormone(FSH) 150IU once a day.
  3. .Ovarian reserve function test abnormalities, including sinus follicle number less than 5-7 AFC or AMH less than 0.5 to 1.1 ng/ml

Ages: 37 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
live birth rate | At birth

SECONDARY OUTCOMES:
cancellation rate | Up to the day of embryo transferred
Pregnancy Rate | Up to 28th day after embryo transferred
abortion rate | Through pregnancy period，average 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China